CLINICAL TRIAL: NCT01935206
Title: Effect of a High-dose Naloxone Infusion on Secondary Hyperalgesia After a First-degree Burn
Brief Title: Effect of High Dose Naloxone on Secondary Hyperalgesia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Manuel Pereira, M.D., Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-2-2012-174
Record Dates: First submitted 2013-08-19; First posted 2013-09-05 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Hyperalgesia; Pain; Naloxone; Opioid Antagonist
Keywords: secondary hyperalgesia; allodynia; mechanical pain threshold; naloxone; endogenous opioids; pain
MeSH Terms: conditions — Hyperalgesia; Pain | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The effect of naloxone (2 mg/kg) on secondary hyperalgesia 168 hours after a first-degree burn-injury is compared to the placebo effect.
  Interventions: Drug: Placebo
- Naloxone (2 mg/kg) (Experimental): The effect of naloxone (2 mg/kg) on secondary hyperalgesia 168 hours after a first-degree burn-injury is compared to the placebo effect.
  Interventions: Drug: Naloxone (2 mg/kg)

INTERVENTIONS:
Drug: Naloxone (2 mg/kg)
  Arms: Naloxone (2 mg/kg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
Recent studies have focused on the role of endogenous opioids on central sensitization. Central sensitization is known to be impaired or altered in chronic pain conditions, as fibromyalgia or chronic tension headache.

Animal studies have shown reinstatement of mechanical hypersensitivity following naloxone administration after resolution of an injury. This suggests latent sensitization.

In the present study, investigators hypothesize that naloxone (2 mg/kg) can reinstate secondary hyperalgesia 168 hours after a first-degree burn-injury. Investigators aim therefore to show that latent sensitization is present in humans and is modulated by endogenous opioids.

ELIGIBILITY:
Inclusion Criteria:

* healthy man
* written informed consent
* ASA 1-2
* BMI 18 < BMI < 30
* normal ultrasound examination of the heart
* normal ECG
* urin sample without traces of opioids

Exclusion Criteria:

* volunteers, who do not understand the Danish language
* participation in another experimental trial in the previous 60 days
* nerve damage or skin lesions in the assessment areas
* neurological or psychiatric condition
* use of psycho-active drugs
* abuse of alcohol or drugs
* chronic pain
* regular use of pain-killers (> 1 a week)
* allergy against morphine or other opioids (including naloxone)
* use of prescription drugs 1 week prior to the trial
* use of over-the-counter medication 48 hours prior to the trial
* urin sample with traces of opioids
* volunteer is not suitable for the trial according to the investigator's consideration

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in Secondary hyperalgesia area (cm2) surrounding a first-degree burn injury before and after infusion of naloxone/placebo | 1h, 2h, 3h, 168h, 168h15min, 168h30min post-burn
  Areas of secondary hyperalgesia surrounding a first degree burn-injury will be assessed before and after infusion of naloxone/placebo.

SECONDARY OUTCOMES:
Change in allodynic area (cm2) surrounding a first-degree burn injury before and after infusion of naloxone/placebo | 1h, 2h, 3h, 168h, 168h15min, 168h30min post-burn
  Areas of allodynia surrounding a first degree burn-injury will be assessed before and after infusion of naloxone/placebo.

OTHER OUTCOMES:
Change in Mechanical Pain Thresholds at primary hyperalgesia site before and after naloxone/placebo infusion | 0h, 168h, 168h30min
  Mechanical Pain Thresholds will be assessed with pinprick stimulators at baseline and after infusion of naloxone/placebo at the primary hyperalgesia site (following a first degree burn) and in the contralateral leg.

CONTACTS AND LOCATIONS:
Overall Officials: Joergen B Dahl, M.D., DMSc, Study Director — Dept Anaesthesiology, HOC, 4231, Rigshospitalet; Mads U. Werner, M.D., Ph.D., DMSc, Principal Investigator — Multidisciplinary Pain Center, 7612, Rigshospitalet, Copenhagen
Locations (2):
- Denmark (2):
  - Dept Anaesthesiology HOC, 4231, Rigshospitalet, Copenhagen, Copenhagen
  - Multidisciplinary Pain Center, Copenhagen, Copenhagen